CLINICAL TRIAL: NCT00054197
Title: CT-2103 vs Gemcitabine or Vinorelbine for the Treatment of PS = 2 Patients With Chemotherapy Naive Advanced Non-Small Cell Lung Cancer (NSCLC): A Phase III Study
Brief Title: Polyglutamate Paclitaxel Compared With Gemcitabine or Vinorelbine in Treating Patients With Advanced or Recurrent Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CTI-PGT304; CDR0000269908 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; paclitaxel poliglumex; Vinorelbine

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: paclitaxel poliglumex
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether polyglutamate paclitaxel is more effective than gemcitabine or vinorelbine in treating non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of polyglutamate paclitaxel with that of gemcitabine or vinorelbine in treating patients who have stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of polyglutamate paclitaxel (CT-2103) vs gemcitabine or vinorelbine, in terms of duration of overall survival, in patients with stage IIIB or IV or recurrent non-small cell lung cancer who have a performance status of 2.
* Compare the safety of these regimens in these patients.
* Compare the disease control (percentage of patients with no disease progression for at least 12 weeks) and time to progression in patients treated with these regimens.
* Compare the response rate in patients with measurable disease treated with these regimens.
* Compare the improvement in lung cancer symptoms in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to gender, disease stage (IV vs other), geographic location (US vs Western Europe and Canada vs the rest of the world), and prior brain metastases (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive polyglutamate paclitaxel (CT-2103) IV over 10 minutes on day 1 every 21 days.
* Arm II: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 every 28 days OR vinorelbine IV over 6-10 minutes on days 1, 8, and 15 every 21 days.

Treatment repeats in both arms for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3 weeks and then every 8 weeks thereafter.

PROJECTED ACCRUAL: A total of 370 patients (185 per treatment arm) will be accrued for this study within 13 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) meeting 1 of the following criteria:

  * Locally advanced or recurrent disease previously treated with radiotherapy and/or surgery
  * Stage IIIB and not a candidate for combined modality therapy
  * Stage IV
* No evidence of small cell carcinoma, carcinoid, or mixed small cell/non-small cell histology
* Cytological diagnosis must be based on the following:

  * No cellular diagnosis by sputum cytology alone
  * Cytologic specimens obtained from brushings, washings, or needle aspiration of a defined lesion or pleural effusion are acceptable
* Measurable or nonmeasurable disease
* Brain metastases allowed provided patient received prior standard antitumor therapy for CNS metastases (e.g., whole brain radiotherapy, stereotactic radioablation, or surgery) and the following conditions are met:

  * Neurologic function stable for at least 2 weeks before study entry
  * Off steroid therapy or on a tapering regimen
  * Recovered from prior therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT/SGPT no greater than 2.5 times ULN (5 times ULN if liver metastases present)
* Alkaline phosphatase no greater than 2.5 times ULN (except for laboratory documentation that demonstrates bone origin)

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No unstable angina
* No myocardial infarction within the past 6 months
* Cardiac conduction abnormalities (e.g., bundle branch block or heart block) allowed provided cardiac status has been stable for at least 6 months prior to study entry

Neurologic

* See Disease Characteristics
* No neuropathy greater than grade 1
* No evidence of unstable neurologic symptoms within the past 4 weeks (2 weeks for neurologic symptoms due to brain metastases)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No intolerance to excipients of polyglutamate paclitaxel (e.g., poly-L-glutamic acid, poloxamer 188, dibasic sodium phosphate, or monobasic sodium hydroxide)
* No clinically significant active infection
* No other concurrent primary malignancy except carcinoma in situ or nonmelanoma skin cancer
* No other unstable medical conditions
* No circumstance that would preclude study completion or follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior systemic biologic agent for lung cancer

Chemotherapy

* See Disease Characteristics
* No prior systemic chemotherapy for lung cancer including radiosensitizing agents

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* Recovered from prior major surgery

Other

* More than 12 weeks since prior participation in any research study or treatment with investigational drugs
* Recovered from prior investigational therapy or stable for 4 weeks before study treatment
* No other concurrent investigational drugs
* No other concurrent systemic antitumor therapy
* No concurrent amifostine
* Concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-01 (Actual); Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghann Smith, Study Chair — PPD, Incorporated
Locations (10):
- United States (10):
  - Cooper Green Hospital, Birmingham, Alabama
  - Medical Oncology/Hematology, Gilroy, California
  - Northwest Oncology and Hematology Associates, Coral Springs, Florida
  - Midwest Cancer Research Group, Incorporated, Skokie, Illinois
  - Medschool Associates North, Reno, Nevada
  - New York Oncology Hematology, P.C. - Latham, Latham, New York
  - Clinical Research Services, Bismarck, North Dakota
  - Charleston Hematology-Oncology, P.A., Charleston, South Carolina
  - Western Washington Medical Group, Everett, Washington
  - Western Washington Oncology, Incorporated, Olympia, Washington

REFERENCES:
- [Result] O'Brien ME, Socinski MA, Popovich AY, Bondarenko IN, Tomova A, Bilynsky BT, Hotko YS, Ganul VL, Kostinsky IY, Eisenfeld AJ, Sandalic L, Oldham FB, Bandstra B, Sandler AB, Singer JW. Randomized phase III trial comparing single-agent paclitaxel Poliglumex (CT-2103, PPX) with single-agent gemcitabine or vinorelbine for the treatment of PS 2 patients with chemotherapy-naive advanced non-small cell lung cancer. J Thorac Oncol. 2008 Jul;3(7):728-34. doi: 10.1097/JTO.0b013e31817c6b68. PMID 18594318